CLINICAL TRIAL: NCT06502795
Title: Quadriceps Strengthening Under Limited Range of Motion Compared to Patient-guided Range of Motion on Pain, Kinesiophobia and Function in Individuals with Patellofemoral Pain: a Randomized Clinical Trial
Brief Title: Quadriceps Strengthening At Different Angles in Patellofemoral Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Gabriel Peixoto Leão Almeida, Principal Investigator, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PFPKarine
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Joint; Chondromalacia Patellae; Physical Therapy Modalities; Quadriceps Muscle; Resistance Training; Exercise Therapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Chondromalacia Patellae

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial with two parallel groups, balanced 1:1 allocation, and double-blind design.
Who Masked: Participant, Investigator
Masking Description: The randomization process will be conducted by a researcher not involved in data collection, using computer-generated random numbers from the Random Allocation Software (version 2.0), in a 1:1 ratio. Randomization codes will be placed in opaque, sequentially numbered envelopes, sealed with a tamper-proof seal, and will be opened only after the envelope has been irreversibly assigned to the participant. The evaluator and the patient will be blinded to the allocation in the experimental and control groups. At the end of the intervention, a masking test will be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Limited Range of Motion Quadriceps Strengthening group (Experimental): The Limited-RoM Quadriceps Strengthening group will perform open-kinetic-chain quadriceps strengthening exercises within a range of 90° to 45° of knee flexion and closed-kinetic-chain within a range of 0° to 45°.
  Interventions: Other: Protected Range Quadriceps Strengthening group
- Patient-Guided Range of Motion Quadriceps Strengthening group (Active Comparator): The Patient-Guided-RoM Quadriceps Strengthening group will perform quadriceps strengthening exercises in both open and closed kinetic chains to the maximum tolerated by the patient based on their symptoms. The patient-guided maximum range of motion will be adjusted based on pain intensity, comfort, and patient response, following a shared decision-making approach with a clinician. The goal will be to maintain exercises at the greatest possible range of motion.
  Interventions: Other: Patient-Guided Range Quadriceps Strengthening group

INTERVENTIONS:
Other: Protected Range Quadriceps Strengthening group — Warm-up: Start with 5 minutes of stationary biking. Then, proceed with two sets of 30-second dynamic stretches targeting the quadriceps, hamstrings, calf muscles, and adductors, followed by static stretching for the abductors.
  Strengthening: Complete 3 sets of 8-12 repetitions for each exercise, aiming for a perceived effort level on the Borg scale between 60% and 80%. Increase the load by 2%-10% when the patient can perform 14 or more repetitions in the final set while maintaining the Borg scale between 60% and 80%.
  For the Leg Extension Machine, maintain a range of motion between 90 to 45 degrees. During Squats and Bulgarian Squats, aim for a range of motion between 0 to 45 degrees.
  Arms: Limited Range of Motion Quadriceps Strengthening group
Other: Patient-Guided Range Quadriceps Strengthening group — Warm-up: 5 minutes of stationary biking. Next, perform two sets of 30-second stretches for the quadriceps, hamstrings, calf muscles, adductors and abductors hip.
  Strengthening: Patients will complete 3 sets of 8 to 12 repetitions for each exercise, aiming for a perceived effort level of 60% to 80% on the Borg scale. Load will be increased by 2% to 10% when patients can complete 14 or more repetitions in the final set while maintaining the Borg scale between 60% and 80%.
  Quadriceps strengthening will be performed at the patient's maximum range guided by symptoms, with pain intensity capped at 5 points on the NPRS. The patient-guided range will be adjusted based on pain intensity, comfort, and patient response, using a shared decision-making approach. The goal is to maintain exercises at the maximum possible range of motion.
  For the Leg Extension Machine, Squats, and Bulgarian Squats, the range of motion will be guided by the patient's pain tolerance.
  Arms: Patient-Guided Range of Motion Quadriceps Strengthening group

SUMMARY:
Introduction: Patellofemoral pain (PFP) is characterized by anterior, retropatellar and/or peripatellar pain during activities such as running, squatting, kneeling, or prolonged sitting. This condition affects approximately 25% of the general population. Given its complex and multifactorial etiology, PFP presents a significant treatment challenge. All clinical practice guidelines recommend strengthening the quadriceps femoris muscle as a key component in the management of PFP. However, exercises aimed at strengthening the quadriceps place considerable stress on the patellofemoral joint and are often poorly tolerated by patients. Clinicians commonly employ a conservative strategy that restricts open kinetic chain knee extension exercises to a limited range of 90° to 45° of knee flexion and closed kinetic chain exercises to 0° to 45°. Yet, restricting the range of motion may result in suboptimal outcomes for patients with higher load tolerance and may foster beliefs regarding knee joint fragility.

Objective: We aim to compare the effects of quadriceps femoris strengthening within a limited range to a patient-guided range of motion on pain, function, knee confidence, and kinesiophobia in individuals with PFP.

Methods: A randomized clinical trial will be conducted with two parallel groups, using a balanced 1:1 allocation and a double-blind design. The study population will include men and women aged 18 to 35 years, diagnosed with PFP. Participants will be randomly assigned to either the limited range group or the patient-guided range of motion group. They will participate in a supervised therapeutic protocol, with sessions averaging 40 minutes, twice a week, for six consecutive weeks. The primary outcome will be pain, assessed using the numerical pain rating scale (0-10), and kinesiophobia, assessed by the Tampa Scale . Secondary outcomes will include pain, self-reported function, measured by the Anterior Knee Pain Scale (AKPS), perceived improvement by the Global Rating of Change Scale, quadriceps strength, kinesiophobia and analgesic consumption.

DETAILED DESCRIPTION:
Participants with patellofemoral pain will be randomized into two intervention groups. All participants will start with a warm-up on a stationary bike, followed by dynamic stretching exercises targeting the quadriceps, hamstrings, calf muscles, adductors, and abductors.

Open kinetic chain exercises will be performed using a leg extension machine, while closed kinetic chain exercises will include free squats and Bulgarian squats.

The Limited-RoM Quadriceps Strengthening group will perform open-kinetic-chain quadriceps strengthening exercises within a range of 90° to 45° of knee flexion and closed-kinetic-chain within a range of 0° to 45°.

The Patient-Guided-RoM Quadriceps Strengthening group will perform quadriceps strengthening exercises in both open and closed kinetic chains to the maximum tolerated by the patient based on their symptoms. The patient-guided maximum range of motion will be adjusted based on pain intensity, comfort, and patient response, following a shared decision-making approach with a clinician. The goal will be to maintain exercises at the greatest possible range of motion.

The identification of the patient-guided angle in both open and closed kinetic chain exercises will be determined as follows: the patient will perform 10 maximum repetitions on the leg with PFP, prioritizing range of motion over load. During the execution, the range of motion and load will be guided by the numerical pain rating scale and the perceived exertion scale.

Participants will complete 12 sessions, twice a week, supervised by a physiotherapist. Assessments will be conducted at baseline, six weeks, and six months, evaluating pain, function, kinesiophobia, crepitus, perception of effect, and weekly pain-killer consumption.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 35 years.
* Diagnosis of patellofemoral pain characterized by peri- or retropatellar pain.
* Pain reproduced in at least two of the following activities: ascending or descending stairs, squatting, kneeling, prolonged sitting, jumping, running, or palpation of the medial and/or lateral facets of the patella.
* Insidious onset of symptoms.
* Symptoms duration of at least three months.
* Minimum score of three on the numerical pain rating scale (NPRS) in the past week.
* Maximum score of 86 points on the Anterior Knee Pain Scale (AKPS)
* In cases of bilateral pain, the more symptomatic knee will be included.

Exclusion Criteria:

* History of surgery and/or fractures in the lower limb joints.
* Other knee joint-related injuries such as meniscal tears, ligament injuries.
* History of patellar subluxation or dislocation.
* Signs of osteoarthritis.
* Patellar and quadriceps tendinopathy.
* Osgood-Schlatter syndrome.
* Presence of knee joint edema.
* Contraindications to resistance exercises informed by a physician.
* Corticosteroid injection within the last 6 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-10-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Knee pain intensity | Knee pain intensity measured by the NPRS after six-week intervention.
  Pain intensity will be measured using the numeric pain rating scale (NPRS), which ranges from 0 to 10 points, where 0 represents no pain and 10 represents the worst possible pain.
Kinesiophobia | Kinesiophobia assessed by the Tampa Scale of Kinesiophobia after six-week intervention.
  The Tampa Scale is a 17-item questionnaire designed to quantify fear of movement and re-injury due to movement and physical activity on a scale from 17 to 68, where 68 indicates higher fear of re-injury due to movement.

SECONDARY OUTCOMES:
Perception of effect | Global Rating of Change Scale after six-week intervention and six-month follow-up.
  Global Rating of Change Scale- This scale consists of 11 points ranging from minus five (extremely worse), zero (no change) to five (completely recovered). For all measures of perceived global effect, participants were asked: "Compared to the beginning of this episode, how would you describe your knee today?" Positive scores indicate better recovery, while negative scores indicate worsening of symptoms.
Knee crepitus | Crepitus during knee extension after six-week intervention.
  The investigator places the palm of their hand over each participant's patella to detect the presence of a grinding sensation during knee extension performed on the leg extension machine. Participants will be instructed to perform two knee extensions as far as they can during the assessment. The test will be considered positive for knee crepitus when a grinding or popping sensation is detected during the range of motion. However, one or two occasional pops will not be considered crepitus. This test has been previously conducted in individuals with PFP.
Weekly analgesic consumption | Weekly, throughout the six-week intervention period.
  The patient will be asked if they have taken pain medications in the last week. If the answer is yes, it will be identified which medications (opioids, anti-inflammatories, or analgesics) were taken and how many medications were consumed.
Knee pain intensity | Knee pain intensity measured by the NPRS at six-month follow-up.
  Pain intensity will be measured using the NPRS, which ranges from 0 to 10 points, where 0 represents no pain and 10 represents the worst possible pain.
Knee function | Self-reported function measured by the AKPS at six-week and six-month follow-up.
  Anterior Knee Pain Scale - AKPS: Specific questionnaire for anterior knee pain comprising 13 items with separate categories related to different levels of knee function.
Kinesiophobia | Kinesiophobia assessed by the Tampa Scale of Kinesiophobia six-month follow-up.
  The Tampa Scale is a 17-item questionnaire designed to quantify fear of movement and re-injury due to movement and physical activity on a scale from 17 to 68, where 68 indicates higher fear of re-injury due to movement.
Quadriceps peak torque | Quadriceps strength measured by the isokinetic dynamometer after six-week intervention.
  Peak torque (Nm) and limb symmetry index on the isokinetic dynamometer, angular velocity of 60 degrees per second, and CON/CON mode.

CONTACTS AND LOCATIONS:
Locations (1):
- Physiotherapy Department, Federal University of Ceará, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Variable characterization will employ descriptive statistical tests (frequency, mean, and standard deviation). Group differences and corresponding confidence intervals will be calculated using mixed linear models incorporating an interaction term for "time versus group." These interaction terms represent group differences (intervention effect). Covariates known to influence clinical outcomes in our study, such as bilateral/unilateral pain presence, symptom duration, and sex, will be incorporated into the statistical models. Statistical analyses will be conducted using SPSS 20.0 for Windows (Statistical Package for the Social Sciences Inc., Chicago, IL, USA) with a significance level set at 5% (α < 0.05).
Supporting Information: SAP

REFERENCES:
- [Background] Almeida GPL, Rodrigues HLDN, Coelho BAL, Rodrigues CAS, Lima POP. Anteromedial versus posterolateral hip musculature strengthening with dose-controlled in women with patellofemoral pain: A randomized controlled trial. Phys Ther Sport. 2021 May;49:149-156. doi: 10.1016/j.ptsp.2021.02.016. Epub 2021 Mar 2. PMID 33689989
- [Background] Collins NJ, Bierma-Zeinstra SM, Crossley KM, van Linschoten RL, Vicenzino B, van Middelkoop M. Prognostic factors for patellofemoral pain: a multicentre observational analysis. Br J Sports Med. 2013 Mar;47(4):227-33. doi: 10.1136/bjsports-2012-091696. Epub 2012 Dec 13. PMID 23242955
- [Background] Collins NJ, Barton CJ, van Middelkoop M, Callaghan MJ, Rathleff MS, Vicenzino BT, Davis IS, Powers CM, Macri EM, Hart HF, de Oliveira Silva D, Crossley KM. 2018 Consensus statement on exercise therapy and physical interventions (orthoses, taping and manual therapy) to treat patellofemoral pain: recommendations from the 5th International Patellofemoral Pain Research Retreat, Gold Coast, Australia, 2017. Br J Sports Med. 2018 Sep;52(18):1170-1178. doi: 10.1136/bjsports-2018-099397. Epub 2018 Jun 20. PMID 29925502
- [Background] Crossley KM, Bennell KL, Cowan SM, Green S. Analysis of outcome measures for persons with patellofemoral pain: which are reliable and valid? Arch Phys Med Rehabil. 2004 May;85(5):815-22. doi: 10.1016/s0003-9993(03)00613-0. PMID 15129407
- [Background] da Cunha RA, Costa LO, Hespanhol Junior LC, Pires RS, Kujala UM, Lopes AD. Translation, cross-cultural adaptation, and clinimetric testing of instruments used to assess patients with patellofemoral pain syndrome in the Brazilian population. J Orthop Sports Phys Ther. 2013 May;43(5):332-9. doi: 10.2519/jospt.2013.4228. Epub 2013 Mar 13. PMID 23485881
- [Background] Escamilla RF, Fleisig GS, Zheng N, Barrentine SW, Wilk KE, Andrews JR. Biomechanics of the knee during closed kinetic chain and open kinetic chain exercises. Med Sci Sports Exerc. 1998 Apr;30(4):556-69. doi: 10.1097/00005768-199804000-00014. PMID 9565938
- [Background] Gallasch CH, Alexandre NM. The measurement of musculoskeletal pain intensity: a comparison of four methods. Rev Gaucha Enferm. 2007 Jun;28(2):260-5. PMID 17907648
- [Background] Giles L, Webster KE, McClelland J, Cook JL. Quadriceps strengthening with and without blood flow restriction in the treatment of patellofemoral pain: a double-blind randomised trial. Br J Sports Med. 2017 Dec;51(23):1688-1694. doi: 10.1136/bjsports-2016-096329. Epub 2017 May 12. PMID 28500081
- [Background] Hansen R, Brushoj C, Rathleff MS, Magnusson SP, Henriksen M. Quadriceps or hip exercises for patellofemoral pain? A randomised controlled equivalence trial. Br J Sports Med. 2023 Oct;57(20):1287-1294. doi: 10.1136/bjsports-2022-106197. Epub 2023 May 3. PMID 37137673
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Lack S, Barton C, Sohan O, Crossley K, Morrissey D. Proximal muscle rehabilitation is effective for patellofemoral pain: a systematic review with meta-analysis. Br J Sports Med. 2015 Nov;49(21):1365-76. doi: 10.1136/bjsports-2015-094723. Epub 2015 Jul 14. PMID 26175019
- [Background] Maclachlan LR, Collins NJ, Matthews MLG, Hodges PW, Vicenzino B. The psychological features of patellofemoral pain: a systematic review. Br J Sports Med. 2017 May;51(9):732-742. doi: 10.1136/bjsports-2016-096705. Epub 2017 Mar 20. PMID 28320733
- [Background] de Oliveira Silva D, Barton C, Crossley K, Waiteman M, Taborda B, Ferreira AS, Azevedo FM. Implications of knee crepitus to the overall clinical presentation of women with and without patellofemoral pain. Phys Ther Sport. 2018 Sep;33:89-95. doi: 10.1016/j.ptsp.2018.07.007. Epub 2018 Jul 17. PMID 30059950
- [Background] de Oliveira Silva D, Barton CJ, Briani RV, Taborda B, Ferreira AS, Pazzinatto MF, Azevedo FM. Kinesiophobia, but not strength is associated with altered movement in women with patellofemoral pain. Gait Posture. 2019 Feb;68:1-5. doi: 10.1016/j.gaitpost.2018.10.033. Epub 2018 Nov 1. PMID 30408709
- [Background] Powers CM, Ho KY, Chen YJ, Souza RB, Farrokhi S. Patellofemoral joint stress during weight-bearing and non-weight-bearing quadriceps exercises. J Orthop Sports Phys Ther. 2014 May;44(5):320-7. doi: 10.2519/jospt.2014.4936. Epub 2014 Mar 27. PMID 24673446
- [Background] Powers CM, Witvrouw E, Davis IS, Crossley KM. Evidence-based framework for a pathomechanical model of patellofemoral pain: 2017 patellofemoral pain consensus statement from the 4th International Patellofemoral Pain Research Retreat, Manchester, UK: part 3. Br J Sports Med. 2017 Dec;51(24):1713-1723. doi: 10.1136/bjsports-2017-098717. Epub 2017 Nov 6. No abstract available. PMID 29109118
- [Background] Priore LB, Azevedo FM, Pazzinatto MF, Ferreira AS, Hart HF, Barton C, de Oliveira Silva D. Influence of kinesiophobia and pain catastrophism on objective function in women with patellofemoral pain. Phys Ther Sport. 2019 Jan;35:116-121. doi: 10.1016/j.ptsp.2018.11.013. Epub 2018 Nov 28. PMID 30529861
- [Background] Smith BE, Selfe J, Thacker D, Hendrick P, Bateman M, Moffatt F, Rathleff MS, Smith TO, Logan P. Incidence and prevalence of patellofemoral pain: A systematic review and meta-analysis. PLoS One. 2018 Jan 11;13(1):e0190892. doi: 10.1371/journal.pone.0190892. eCollection 2018. PMID 29324820
- [Background] Stathopulu E, Baildam E. Anterior knee pain: a long-term follow-up. Rheumatology (Oxford). 2003 Feb;42(2):380-2. doi: 10.1093/rheumatology/keg093. PMID 12595641
- [Background] Steinkamp LA, Dillingham MF, Markel MD, Hill JA, Kaufman KR. Biomechanical considerations in patellofemoral joint rehabilitation. Am J Sports Med. 1993 May-Jun;21(3):438-44. doi: 10.1177/036354659302100319. PMID 8346760
- [Background] Willy RW, Hoglund LT, Barton CJ, Bolgla LA, Scalzitti DA, Logerstedt DS, Lynch AD, Snyder-Mackler L, McDonough CM. Patellofemoral Pain. J Orthop Sports Phys Ther. 2019 Sep;49(9):CPG1-CPG95. doi: 10.2519/jospt.2019.0302. PMID 31475628